CLINICAL TRIAL: NCT04436978
Title: What is the Optimal Antithrombotic Strategy in Patients With Atrial Fibrillation Having Acute Coronary Syndrome or Undergoing Percutaneous Coronary Intervention?
Brief Title: What is the Optimal Antithrombotic Strategy in Patients With Atrial Fibrillation Undergoing PCI?
Acronym: WOEST-3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Professor dr., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL81102.100.22; 2022-001298-30 (EudraCT Number)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Atrial Fibrillation; Atrial Flutter; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Bleeding; Stroke; Stent Thrombosis; Embolism; Coronary Artery Disease
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Atrial Fibrillation; Atrial Flutter; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Oral Anticoagulant; NOAC - Novel Oral Anticoagulant; DOAC - Direct Oral Anticoagulant; DAPT - Dual Antiplatelet Therapy; Antithrombotic Therapy; Dual Therapy; Triple Therapy; Bleeding; Thrombosis; Stroke; Stent Thrombosis; Systemic Embolism; Percutaneous coronary intervention; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Atrial Fibrillation; Atrial Flutter; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Hemorrhage; Stroke; Embolism; Coronary Artery Disease; Thrombosis | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Intervention Model Description: The study is designed as a multicentre open label randomized controlled superiority trial with regards to safety and non-inferiority trial with regards to efficacy.
  Participating study centres will enrol patients undergoing PCI who have previously or newly diagnosed AF and indication for NOAC. As soon as possible, but within 72 hours after PCI, patients will be randomized 1:1 to either
  * 30 days DAPT (asprin + P2Y12 inhibitor), followed by guideline-directed therapy (edoxaban + P2Y12 inhibitor)
  * Standard guideline-directed therapy (edoxaban + P2Y12 inhibitor, aspirin limited to in-hospital use or up to 30 days in selected high-risk patients)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First month DAPT (Active Comparator): 30-day DAPT (aspirin + P2Y12 inhibitor). After 30 days all patients will be treated with edoxaban and P2Y12 inhibitor.
  Selection of P2Y12 inhibitor is at the discretion of the treating physician, depending on both bleeding and ischemic risk. Dosage of aspirin and P2Y12 inhibitor is according to local guidelines.
  NOAC of choice will be edoxaban. Patients will be treated with the recommended dose of 60mg once daily or the reduced dose of 30mg once daily.
  Interventions: Drug: 30-day DAPT
- Guideline-directed therapy (Active Comparator): Standard guideline-directed therapy (edoxaban + P2Y12 inhibitor, aspirin limited to in-hospital use or up to 30 days in selected high-risk patients). After 30 days all patients will be treated with edoxaban and P2Y12 inhibitor.
  Selection of P2Y12 inhibitor is at the discretion of the treating physician, depending on both bleeding and ischemic risk. Dosage of aspirin and P2Y12 inhibitor is according to local guidelines.
  NOAC of choice will be edoxaban. Patients will be treated with the recommended dose of 60mg once daily or the reduced dose of 30mg once daily.
  Interventions: Drug: Guideline-directed therapy

INTERVENTIONS:
Drug: 30-day DAPT — DAPT (aspirin + P2Y12 inhibitor) during the first 30 days following PCI. After 30 days, all patients will be treated with edoxaban and a P2Y12 inhibitor.
  Arms: First month DAPT
Drug: Guideline-directed therapy — Guideline-directed therapy (edoxaban + P2Y12 inhibitor, aspirin limited to in-hospital use or up to 30 days in selected high-risk patients)
  Arms: Guideline-directed therapy

SUMMARY:
The optimal antithrombotic management in patients with coronary artery disease (CAD) and concomitant atrial fibrillation (AF) is unknown. AF patients are treated with oral anticoagulation (OAC) to prevent ischemic stroke and systemic embolism and patients undergoing percutaneous coronary intervention (PCI) are treated with dual antiplatelet therapy (DAPT), i.e. aspirin plus P2Y12 inhibitor, to prevent stent thrombosis (ST) and myocardial infarction (MI). Patients with AF undergoing PCI were traditionally treated with triple antithrombotic therapy (TAT, i.e. OAC plus aspirin and P2Y12 inhibitor) to prevent ischemic complications. However, TAT doubles or even triples the risk of major bleeding complications. More recently, several clinical studies demonstrated that omitting aspirin, a strategy known as dual antithrombotic therapy (DAT) is safer compared to TAT with comparable efficacy.

However, pooled evidence from recent meta-analyses suggests that patients treated with DAT are at increased risk of MI and ST. Insights from the AUGUSTUS trial showed that aspirin added to OAC and clopidogrel for 30 days, but not thereafter, resulted in fewer severe ischemic events. This finding emphasizes the relevance of early aspirin administration on ischemic benefit, also reflected in the current ESC guideline. However, because we consider the bleeding risk of TAT unacceptably high, we propose to use a short course of DAPT (omitting OAC for 1 month). There is evidence from the BRIDGE study that a short period of omitting OAC is safe in patients with AF. In this study, these patients are treated with DAPT, which also prevents stroke, albeit not as effective as OAC. This temporary interruption of OAC will allow aspirin treatment in the first month post-PCI where the risk of both bleeding and stent thrombosis is greatest.

The WOEST 3 trial is a multicentre, open-label, randomised controlled trial investigating the safety and efficacy of one month DAPT compared to guideline-directed therapy consisting of OAC and P2Y12 inhibitor combined with aspirin up to 30 days. We hypothesise that the use of short course DAPT is superior in bleeding and non-inferior in preventing ischemic events. The primary safety endpoint is major or clinically relevant non-major bleeding as defined by the ISTH at 6 weeks after PCI. The primary efficacy endpoint is a composite of all-cause death, myocardial infarction, stroke, systemic embolism, or stent thrombosis at 6 weeks after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. Undergoing successful PCI (either ACS or elective PCI)
3. History of or newly diagnosed (<72 hours after PCI/ACS) atrial fibrillation or flutter with a long-term (≥ 1 year) indication for OAC

Exclusion Criteria:

1. Contra indication to edoxaban, aspirin or all P2Y12 inhibitors
2. Current indication for OAC besides atrial fibrillation/flutter (e.g. venous thromboembolism)
3. <12 months after any stroke
4. CHADSVASc score ≥7
5. Moderate to severe mitral valve stenosis (AVA ≤1.5 cm2)
6. Mechanical heart valve prosthesis
7. Intracardiac thrombus or apical aneurysm requiring OAC
8. Poor LV function (LVEF <30%) with proven slow-flow
9. History of intracranial haemorrhage
10. Active bleeding on randomization
11. History of intraocular, spinal, retroperitoneal, or traumatic intra-articular bleeding, unless the causative factor has been permanently resolved
12. Recent (<1 month) gastrointestinal haemorrhage, unless the causative factor has been permanently resolved.
13. Known coagulopathy
14. Severe anaemia requiring blood transfusion or thrombocytopenia <50 × 109/L
15. BMI >40 or bariatric surgery
16. Kidney failure (eGFR <15)
17. Active liver disease (ALT, ASP, AP >3x ULN or active hepatitis A, B or C)
18. Active malignancy excluding non-melanoma skin cancer
19. Life expectancy <1 year
20. Pregnancy or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | 6 weeks
  Major or clinically relevant non-major bleeding as defined by the International Society of Thrombosis and Haemostasis
Primary efficacy endpoint | 6 weeks
  Composite of all-cause death, myocardial infarction, stroke, systemic embolism, or stent thrombosis

SECONDARY OUTCOMES:
Bleeding complications | 6 months
  Major or clinically relevant non-major bleeding as defined by the International Society of Thrombosis and Haemostasis
Thrombotic complications | 6 months
  Composite of all-cause death, myocardial infarction, stroke, systemic embolism, or stent thrombosis
Net clinical benefit | 6 weeks, 3 months, 6 months
  Composite of major bleeding, myocardial infarction, stroke, systemic embolism all-cause death and stent thrombosis
Clinical symptom severity | 6 weeks, 3 months, 6 months
  CCS grade
All-cause death | 6 weeks, 3 months, 6 months
  All-cause death as defined by ARC-2 and SCTI
Myocardial infarction | 6 weeks, 3 months, 6 months
  Myocardial infarction as defined by the 4th Universal Definition of Myocardial Infarction
Stroke | 6 weeks, 3 months, 6 months
  Stroke as defined by VARC-2 definitions
Systemic embolism | 6 weeks, 3 months, 6 months
  Systemic embolism according to ENTRUST-AF PCI definition
Stent thrombosis | 6 weeks, 3 months, 6 months
  Stent thrombosis as defined by ARC-2
Major bleeding | 6 weeks, 3 months, 6 months
  Major bleeding as defined by BARC 3 or 5
Clinically relevant non-major bleeding | 6 weeks, 3 months, 6 months
  CRNM as defined by BARC 2

OTHER OUTCOMES:
Quality of life as assessed by the EuroQol-5D-5L questionnaire | 6 weeks, 3 months, 6 months
  EuroQol-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën M ten Berg, Prof, MD, Principal Investigator — St. Antonius Hospital
Locations (20):
- Belgium (10):
  - ASZ Aalst, Aalst
  - UZ Antwerpen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria Middelares Gent, Ghent
  - Jan Yperman, Ieper
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Netherlands (10):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Treant Zorggroep, Emmen
  - Zuyderland Ziekenhuis, Heerlen
  - Tergooi MC, Hilversum
  - St. Antonius Hospital, Nieuwegein
  - Hagaziekenhuis, The Hague
  - Elisabeth Tweesteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: Yes
Will individual participant data be available? Yes
  What data in particular will be shared? Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  What other documents will be available? Study Protocol, informed consent form, clinical study report
  When will data be available (start and end dates)? Within 1 year following article publication. End date to be determined.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? To achieve aims in the approved proposal.
  By what mechanism will data be made available? Proposals should be directed to as.verburg@antoniusziekenhuis.nl. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within 1 year following article publication. End date to be determined.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Verburg A, Bor WL, Kucuk IT, Henriques JPS, Vink MA, Ruifrok WT, Plomp J, Heestermans TACM, Schotborgh CE, Vlaar PJ, Magro M, Rikken SAOF, van den Broek WWA, van Mieghem CAG, Cornelis K, Rosseel L, Dujardin KS, Vandeloo B, Vandendriessche T, Ferdinande B, van 't Hof AWJ, Tijssen JGP, Limbruno U, De Caterina R, Rubboli A, Angiolillo DJ, Adriaenssens T, Dewilde W, Ten Berg JM. Temporary omission of oral anticoagulation in atrial fibrillation patients undergoing percutaneous coronary intervention: rationale and design of the WOEST-3 randomised trial. EuroIntervention. 2024 Jul 15;20(14):e898-e904. doi: 10.4244/EIJ-D-24-00100. PMID 39007830